CLINICAL TRIAL: NCT05314634
Title: The Effect of Acute Concurrent Exercise on Executive Function: An Event-Related Potential Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Professor, National Taiwan Normal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACNL_rueihongli_CE
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Executive Function
Keywords: acute exercise; concurrent exercise; cognitive flexibility
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to three group, namely the concurrent exercise group (CE), the aerobic exercise group (AE), and the reading control group (RC). Participants in CE groups were asked to finish 5 min warm-up, 12 min aerobic exercise, 13 min resistance exercise, and 5 min cool down. Participants in the AE group were asked to finish 5 min warm-up, 25 min aerobic exercise, and 5 min cool down. Participants in RC group were required to finish 35 min reading. All groups took a 30 min cognitive test before and after the intervention. The blood lactate were collected before, 17 minutes after, and after the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- concurrent exercise group, CE (Experimental): Participants conduct 5-min warm up, 12-min aerobic exercise, 13-min resistance exercise, and 5-min cool down.
  Interventions: Behavioral: concurrent exercise
- aerobic exercise group, AE (Experimental): Participants conduct 5-min warm up, 25-min aerobic exercise, and 5-min cool down.
  Interventions: Behavioral: aerobic exercise
- reading control group, RC (No Intervention): Participants conduct reading for 35 minutes.

INTERVENTIONS:
Behavioral: concurrent exercise — Participants conduct warm up for 5-min, aerobic exercise for 12-min, resistance exercise for 13-min, and 5-min cool down.
  Arms: concurrent exercise group, CE
Behavioral: aerobic exercise — Participants conduct warm up for 5-min, resistance training for 25-min, and 5-min cool down.
  Arms: aerobic exercise group, AE

SUMMARY:
Executive function is a high-level cognition which plays an important role in our life. Meta-analysis study has demonstrated that acute exercise could improve executive function. However, it is still unclear whether executive function can be enhanced by the concurrent exercise that combines aerobic and resistance exercise. Moreover, previous studies indicated that acute exercise could increase the concentration of blood lactate which is positive correlated to executive function. It is still unclear whether the effect of acute concurrent exercise on executive function is mediated by blood lactate. Therefore, the purposes of present study are: (1) Measuring the effect of acute concurrent exercise and aerobic exercise on executive function. (2) Measuring whether the effect of acute concurrent exercise on executive function is mediated by blood lactate.

DETAILED DESCRIPTION:
Executive function is a high-level cognition which plays an important role in academic performance, career, and interpersonal relationship. Meta-analysis study has demonstrated that acute exercise could improve executive function, and also observed similar positive effect through both aerobic and resistance exercise. However, it is still unclear whether executive function can be enhanced by the concurrent exercise that combines aerobic and resistance exercise. Moreover, previous studies indicated that acute exercise could increase the concentration of blood lactate which is positive correlated to executive function. It is still unclear whether the effect of acute concurrent exercise on executive function is mediated by blood lactate. Therefore, the purposes of present study are: (1) Measuring the effect of acute concurrent exercise and aerobic exercise on executive function. (2) Measuring whether the effect of acute concurrent exercise on executive function is mediated by blood lactate.

ELIGIBILITY:
Inclusion Criteria:

1. no history of psychiatric or neurological disorders
2. no history of cardiovascular disease
3. normal or corrected to normal vision and normal color perception
4. right handed
5. 18.5 < BMI < 27

Exclusion Criteria:

1. Diagnosed with epilepsy

Ages: 21 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Ph.D., Study Director — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Concurrent Exercise Group, CE | Aerobic Exercise Group, AE | Reading Control Group, RC
Started | 26 | 26 | 26
Completed | 26 | 26 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concurrent Exercise Group, CE | Aerobic Exercise Group, AE | Reading Control Group, RC | Total
Number analyzed (Participants) | 26 | 26 | 26 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 26 | 78
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.81 (2.00) | 22.85 (1.54) | 22.81 (1.90) | 22.82 (1.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 13 | 40
  Male | 12 | 13 | 13 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 26 | 26 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 26 | 26 | 26 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 26 | 26 | 26 | 78
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.25 (2.02) | 20.42 (2.42) | 21.72 (1.82) | 21.13 (2.14)

OUTCOME MEASURES:

1. Primary Outcome: Task Switch Test Response Times
Description: The shifting aspect of executive function was assessed using a computerised task-switching test. Each participant (N=78) completed 384 trials across six blocks (64 trials per block). The test consisted of two types of cognitive tasks: (1) number magnitude judgment (greater/less than 5) for digits 1-9 presented in solid-line squares, and (2) odd/even judgment for numbers presented in dotted-line squares. Performance was analysed by calculating each participant's mean response time (milliseconds) under four conditions:
  Homogeneous condition: Blocks where participants performed the same task repeatedly (Blocks 1 & 2, e.g., AAAA or BBBB) Heterogeneous condition: Blocks where tasks were mixed (Blocks 3-6, e.g., AABBAA) Non-switch trials: Consecutive trials of the same task type within heterogeneous blocks (e.g., AA or BB) Switch trials: Trials where the task changed from the previous trial within heterogeneous blocks (e.g., AB or BA) Lower response time represents better task perform
Time Frame: 30 minutes
Population: The analysis was based on participants' mean response times under four cognitive conditions (Homogeneous, Heterogeneous, Non-switch, and Switch), derived from their performance across 384 trials (6 blocks × 64 trials).
Measure: Mean (Standard Error); unit: millisecond
Units Other Than Participants: trials
Arm/Group | Concurrent Exercise Group, CE | Aerobic Exercise Group, AE | Reading Control Group, RC
Number analyzed (Participants) | 26 | 26 | 26
Number analyzed (trials) | 384 | 384 | 384
millisecond
  Heterogeneous: number analyzed (trials) | 256 | 256 | 256
  Heterogeneous | 783.97 (11.65) | 788.76 (11.66) | 839.46 (11.65)
  Homogeneous: number analyzed (trials) | 128 | 128 | 128
  Homogeneous | 566.46 (14.67) | 547.82 (14.70) | 618.30 (14.72)
  Non-switch: number analyzed (trials) | 128 | 128 | 128
  Non-switch | 737.73 (11.63) | 753.98 (11.62) | 797.48 (11.62)
  Switch: number analyzed (trials) | 128 | 128 | 128
  Switch | 833.32 (13.34) | 825.39 (13.34) | 882.18 (13.34)

2. Other Pre Specified Outcome: Blood Lactate
Description: The lactic acid system is one of the important systems of human energy metabolism. In addition to supplying energy to muscles, it can also be used as an energy source for brain energy metabolism. When people doing exercise, the concentration of blood lactate will be increased, and the lactate acid system will replace the glucose system as the main energy source for the brain. In the present study, blood lactate were collected from fingertip with a lancet and measured by lactate analyzer before, 17 minutes after, and after intervention.
Time Frame: before intervention, 17 minutes after intervention, and immediately after the 35 minute intervention
Population: Blood lactate samples were collected from fingertip with a lancet and measured by lactate analyzer at three time points: before, 17 minutes after, and after intervention (three blood samples were collected from each participant).
Measure: Mean (Standard Error); unit: mmol/l
Arm/Group | Concurrent Exercise Group, CE | Aerobic Exercise Group, AE | Reading Control Group, RC
Number analyzed (Participants) | 26 | 26 | 26
mmol/l
  Before intervention | 2.95 (0.32) | 3.09 (0.32) | 2.4 (0.32)
  Seventeen minutes after intervention | 5.58 (0.41) | 5.27 (0.41) | 2.13 (0.41)
  After intervention | 8.94 (0.44) | 4.65 (0.44) | 2.44 (0.44)

3. Other Pre Specified Outcome: Stroop Task
Description: The Stroop task consists of neutral, congruent, and incongruent trials. In neutral trials, colored rectangles were presented and participants were instructed to respond to whether the squares were red, blue, or green. For congruent and incongruent trials, participants were presented with the names of the three Chinese color words of 紅 (red), 藍 (blue), or 綠 (green) printed in either the same (congruent) or different (incongruent) ink color and instructed to respond to the color of the ink while inhibiting the meaning of the word.
Time Frame: 30 minutes
Population: Given temporal constraints, the Stroop task was not measured in this study.
Arm/Group | Concurrent Exercise Group, CE | Aerobic Exercise Group, AE | Reading Control Group, RC
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year.
Arm/Group | Concurrent Exercise Group, CE | Aerobic Exercise Group, AE | Reading Control Group, RC
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT05314634/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT05314634/SAP_001.pdf